CLINICAL TRIAL: NCT01115517
Title: A Pilot Study to Assess Safety and Efficacy of Intraoperative Topical Mitomycin C and Bevacizumab (Avastin) Applied to Bare Sclera in Pterygium Surgery
Brief Title: Safety Study of Avastin Used as Adjunctive Therapy in Pterygium Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Hermann Eye Center (Other)
Responsible Party: Principal Investigator, Nan Wang, Clinical Associate Professor - Ophthalmology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pterygium Avastin study
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2016-09-02 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Bevacizumab; Mitomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab
- Mitomycin C (Active Comparator)
  Interventions: Drug: Mitomycin C

INTERVENTIONS:
Drug: Bevacizumab — 1.25 mg/mL applied one time intraoperatively using bevacizumab-soaked filter paper manually applied to bare sclera during pterygium surgery for 2 minutes, followed by copious rinsing with balanced salt solution.
  Other Names: Bevacizumab (Avastin)
  Arms: Bevacizumab
Drug: Mitomycin C — Mitomycin C 0.02% will be applied to bare sclera during pterygium surgery using a medication-soaked filter paper for a duration of two minutes. After medication administration, the ocular surface will be copiously irrigated with balanced salt solution.
  Arms: Mitomycin C

SUMMARY:
This study will evaluate the efficacy and safety of the use of bevacizumab (Avastin) as an adjunctive medication during pterygium surgery in preventing pterygium recurrence. A pterygium is a white fleshy growth on the surface of the eye, which can be removed surgically. However, after surgical removal, pterygia can recur. One way of minimizing recurrence is by applying a medication called mitomycin C to the surface of the eye during pterygium surgery. However, mitomycin is associated with certain side effects, such as thinning of the eye wall and poor wound healing. Bevacizumab has a different mechanism of action and there is some evidence that it may be useful in preventing pterygium recurrence. In this study, the safety and efficacy of adjunctive intraoperative use of bevacizumab and mitomycin C for preventing pterygium recurrence will be directly compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Presence of primary or recurrent pterygium
* Pterygium grows greater than 2mm onto cornea from limbus (using slit lamp light beam to measure size)
* Pterygium is inducing astigmatism greater than 1 diopter compared to the fellow eye (to be determined by automated keratometry and manifest refraction)
* The pterygium is symptomatic (irritation, inflammation, strabismus, decreased visual acuity)

Exclusion Criteria:

* Age less than 18
* Age greater than 80
* Any systemic rheumatologic or autoimmune disorder (autoimmune hepatitis, bullous pemphigoid, celiac disease, Crohn's disease, dermatomyositis, Graves' disease, Hashimoto's thyroiditis, systemic lupus erythematosus, mixed connective tissue disease, pemphigus vulgaris, psoriasis, polymyositis, rheumatoid arthritis, scleroderma, Sjogren's disease, ulcerative colitis, vasculitis, Wegener's granulomatosus)
* Women who are potentially child-bearing (no possibility of pregnancy for at least one month after surgery)
* Any use within the past two months of topical eye drops other than artificial tears in the study eye
* Any previous intravitreal injections of any medication in the study eye
* Any previous use of systemic, topical, or intravitreal bevacizumab in either eye
* Any history of subconjunctival injections in the study eye within the past year
* Any history of scleral or corneal laceration in the study eye
* Ocular surgery within the past 3 months in the study eye
* History of scleral buckle placement in the study eye
* History of glaucoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nan Wang, MD, PhD, Principal Investigator — University of Texas at Houston Health Science Center, Robert Cizik Eye Clinic
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - Robert Cizik Eye Clinic, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 participants were consented and screened for this study, however only 39 of the 51 met eligibility criteria and were randomized.
Period: Overall Study
Arm/Group | Bevacizumab | Mitomycin C
Started | 18 | 21
Completed | 14 | 16
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Mitomycin C | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11) | 43.9 (9.4) | 49.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Recurrence of Pterygia up to 1 Year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Bevacizumab | Mitomycin C
Number analyzed (Participants) | 14 | 16
participants | 0 | 3

2. Secondary Outcome: Number of Participants Who Had Complications From the Time of Treatment to Recurrence
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Bevacizumab | Mitomycin C
Number analyzed (Participants) | 14 | 16
participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Had Related Serious Adverse Events From the Time of Treatment to 1 Year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Bevacizumab | Mitomycin C
Number analyzed (Participants) | 14 | 16
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Potentially related adverse events and serious adverse events were collected and analyzed from the time of treatment to the end of study.
Arm/Group | Bevacizumab | Mitomycin C
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No